CLINICAL TRIAL: NCT03614533
Title: A Phase 2 Randomized, Double-Blind, Controlled Trial of the Safety and Immunogenicity of Typhoid Conjugate Vaccine (Vi-TCV) Among Children Younger Than 2 Years in Ouagadougou, Burkina Faso
Brief Title: Typhoid Conjugate Vaccine Trial Among Children Younger Than 2 Years in Ouagadougou, Burkina Faso
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Groupe de Recherche Action en Sante (Other)
Responsible Party: Principal Investigator, Matthew Laurens, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HP-00081030
Record Dates: First submitted 2018-07-11; First posted 2018-08-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Typhoid
Keywords: Typhoid in Burkina Faso; Typhoid Conjugate Vaccine
MeSH Terms: conditions — Typhoid Fever | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vi-Typhoid Conjugate Vaccine (Vi-TCV) (Experimental): Children will receive a single 0.5-ml dose of Vi-TCV administered by the intramuscular route.
  Interventions: Biological: Vi-Typhoid Conjugate Vaccine (Vi-TCV)
- Inactivated Poliovirus Vaccine (IPV) (Active Comparator): Children will receive a single 0.5-ml dose of Inactivated Poliovirus Vaccine (IPV) by the intramuscular route.
  Interventions: Biological: Inactivated Poliovirus Vaccine (IPV)

INTERVENTIONS:
Biological: Vi-Typhoid Conjugate Vaccine (Vi-TCV) — Single 0.5-ml intramuscular injection
  Arms: Vi-Typhoid Conjugate Vaccine (Vi-TCV)
Biological: Inactivated Poliovirus Vaccine (IPV) — Single 0.5-ml intramuscular injection
  Arms: Inactivated Poliovirus Vaccine (IPV)

SUMMARY:
Typhoid fever is an illness that may cause mild effects in children, such as fever and feeling tired, or it may cause serious effects-- even death. A new typhoid vaccine has recently been recommended by the World Health Organization (WHO) to prevent typhoid in children. But this new typhoid vaccine has not been tested with all of the vaccines given to children in Burkina Faso. The investigators want to look at this new vaccine, and study how safe it is in children in Burkina Faso and how their immune systems respond to the vaccine when given with other vaccines, such as yellow fever and meningitis A vaccines.

The investigators plan to vaccinate 100 children between the ages of 9-11 months, and 150 children between the ages of 15 months and 2 years, in Ouagadougou, Burkina Faso, with either the typhoid vaccine or a vaccine against another illness called polio.

Children will have follow-up visits on days 3, 7, 28 and 180. One teaspoon of blood will be collected on days 0 and 28.

DETAILED DESCRIPTION:
This study will be divided into two cohorts, by age, with separate study designs. The first cohort will include children 9 through 11 months of age. The second cohort will comprise children 15 through 23 months of age. The purpose of this detailed evaluation of safety and immunogenicity is to assess the reactogenicity of the vaccine and the immune responses to Vi-TCV. Serum specimens will be collected from all participants on study day 0 (before vaccination) and on post-vaccination study day 28 to quantify anti-Vi and anti-tetanus toxoid antibodies. All children will have an additional 0.5 mL of blood collected on study day 0 before study vaccination to test for the presence of malaria parasitemia at baseline.

Children 9 through 11 months of age in the Ouagadougou study area will be eligible for the first age cohort, which will be a double-blind, individually randomized, controlled trial. Up to 100 children in this cohort will be randomized in a 1:1 ratio to receive Vi-TCV (Group 1) or IPV (Group 2). Participants will be unaware of which study vaccine, Vi-TCV or IPV, is received. Vi-TCV or IPV will be administered with measles-rubella vaccine (MR) and YFV, as per Burkina Faso Expanded Programme on Immunization (EPI) schedule. These 9 through 11-month-old children will have immunogenicity to Vi-TCV, YFV, and tetanus toxoid assessed on study days 0 and 28.

Children 15 through 23 months of age in the Ouagadougou study area will be eligible for the second cohort, a randomized study of the safety and immunogenicity of Vi-TCV when co-administered with routine Expanded Programme on Immunisation (EPI) vaccines (MAV and MR) or given alone, and MAV immunogenicity when co-adminstered or given alone. Participants in this cohort (up to 150) will be randomized 1:1:1 to one of three treatment groups, as follows. The first group of participants (Group A) will receive Vi-TCV and IPV at study day 0, with a subsequent dose of MAV at study day 28; the second group of participants (Group B) will receive MAV and Vi-TCV at study day 0; the third group (Group C) will receive MAV and IPV at study day 0. All children will receive MR at study day 0. Cohort 1 will be unblinded on day 28 for safety and follow-up and to ensure MAV receipt in Group A. These 15 through 23-month-old children will have antibody to meningococcal A vaccine, anti-Vi antibody, and tetanus toxoid antibody assessed on study days 0 and 28.

Participants in both cohorts will have home or clinic visits on days 3 and 7 following vaccination for solicitation of local and systemic adverse events. Non-serious adverse events will be assessed up until the study day 28 visit. Serious adverse events will be captured throughout study follow-up and actively during the study day 180 visit.

ELIGIBILITY:
Inclusion Criteria: Each subject receiving study vaccine (Vi-TCV or IPV) must satisfy the following inclusion criteria at study entry:

* Male or female child 9 through11 months of age for cohort 1, or 15 months through 23 months of age for cohort 2, and in good health at the time of study vaccination.
* A child whose parent or guardian resides primarily within the study area at the time of study vaccinations and who intends to be present in the area for the duration of the trial.
* A child whose parent or guardian has voluntarily given informed consent.

Exclusion Criteria: No subject receiving study vaccine (Vi-TCV or IPV) may have any of the following exclusion criteria at study entry:

* History of documented hypersensitivity to any component of the vaccine.
* Prior receipt of any typhoid vaccine.
* History of severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis.
* Known history of diabetes, tuberculosis, cancer, chronic kidney, heart, or liver disease, progressive neurological disorders, poorly controlled seizures, or terminal illness.
* Severe malnutrition as determined by a MUAC < 12.5 cm.
* Receipt of any other investigational intervention in the last 6 months or anticipated during the course of the study.
* Receipt of blood products in the last 6 months.
* Known HIV infection or exposure or other immunosuppressive conditions.
* Receipt of systemic immunosuppressant or systemic corticosteroids.
* Receipt of any measles-rubella-containing vaccine for children younger than 1 year of age.
* Any condition determined by the investigator likely to interfere with evaluation of the vaccine or to be a significant potential health risk to the child or make it unlikely that the child would complete the study.

Temporary Exclusion Criteria: The following will be considered a temporary contraindication to enrollment and vaccination. If this applies, the participant will be temporarily excluded for vaccination until 48 hours has passed. A re-assessment will be needed to ensure the temporary exclusion criteria no longer exist:

• Reported fever within 24 hours before vaccination.

An additional temporary exclusion criteria for cohort 2 will be:

• Receipt of measles-rubella vaccine in the one month before enrollment, as determined by parental history or vaccination card. A child may be reassessed after 30 days has passed since receipt of MR vaccine.

Ages: 9 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Safety of Vi-TCV After 7 Days | Within 7 days after vaccination
  The proportion of participants who develop adverse events detected in the first 7 days after vaccination.
Safety of Vi-TCV After 6 Months | Within 6 months after vaccination
  The proportion of participants who experience serious adverse events within 6 months of vaccination in all participants.
Safety of Vi-TCV After 28 Days | Within 28 days after vaccination
  The proportion of participants who experience other non-serious adverse events up to 28 days following vaccination, in a subset of participants.

SECONDARY OUTCOMES:
Noninterference Vi-TCV with Yellow Fever Vaccine | At days 0 and 28
  The immunogenicity of YF when given with and without Vi-TCV, measured by yellow fever plaque reduction neutralization test at study days 0 and 28 among children in cohort 1, groups 1 and 2.
Noninterference of Vi-TCV with Meningitis A Vaccine | At days 0 and 28
  The immunogenicity of MAV when given with and without Vi-TCV, measured by serum bactericidal antibody at study days 0 and 28 among children in cohort 2, groups 4 and 5.
Noninterference of Yellow Fever Vaccine with Vi-TCV | At days 0 and 28
  The immunogenicity of Vi-TCV when given with YF, measured by ELISA for anti-Vi percent seroconversion (>4-fold increase in geometric mean titer (GMT)) and GMT at study days 0 and 28 among children in cohort 1, groups 1 and 2.
Noninterference of Meningitis A Vaccine with Vi-TCV | At days 0 and 28
  The immunogenicity of Vi-TCV when given with and without MAV, measured by ELISA for anti-Vi percent seroconversion (>4-fold increase in GMT) and GMT at study days 0 and 28 among children in cohort 2, groups 3 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Laurens Matthew, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Groupe de Recherche Action en Santé (GRAS), Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laurens MB, Sirima SB, Rotrosen ET, Siribie M, Tiono A, Ouedraogo A, Liang Y, Jamka LP, Kotloff KL, Neuzil KM. A Phase II, Randomized, Double-blind, Controlled Safety and Immunogenicity Trial of Typhoid Conjugate Vaccine in Children Under 2 Years of Age in Ouagadougou, Burkina Faso: A Methods Paper. Clin Infect Dis. 2019 Mar 7;68(Suppl 2):S59-S66. doi: 10.1093/cid/ciy1104. PMID 30845330